CLINICAL TRIAL: NCT01885104
Title: Evaluation of Oral Tolerance MiraLAX Solution Concentrate in Subjects With Chronic Constipation
Brief Title: Safety and Tolerability of Oral Polyethylene Glycol (PEG 3350) Solution in Participants With Constipation (MK-8114-003)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18127; CL2012-13 (Other: Consumer Health Protocol Number); 8114-003 (Other: Merck)
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Polyethylene Glycols; polyethylene glycol 3350

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG 3350 (Experimental): Participants will receive a 17 g dose of PEG 3350 solution concentrate in a volume of approximately 30 mL, once a day, for 14 days. Bisacodyl laxative tablets, 5.0 mg, 1 to 3 tablets in a single daily dose, will be provided for use as a rescue medication if a participant has not had a bowel movement for 72 hours after start of treatment.
  Interventions: Drug: Polyethylene Glycol (PEG 3350); Drug: Bisacodyl laxative tablets (rescue medication)
- Placebo (Placebo Comparator): Participants will receive a 17 g dose of Placebo solution concentrate in a volume of approximately 30 mL, once a day, for 14 days. Bisacodyl laxative tablets, 5.0 mg, 1 to 3 tablets in a single daily dose, will be provided for use as a rescue medication if a participant has not had a bowel movement for 72 hours after start of treatment.
  Interventions: Drug: Placebo; Drug: Bisacodyl laxative tablets (rescue medication)

INTERVENTIONS:
Drug: Polyethylene Glycol (PEG 3350) — Oral 17 g dose of PEG 3350 solution concentrate in a volume of approximately 30 mL, once a day, for 14 days.
  Other Names: MiraLAX Solution Concentrate
  Arms: PEG 3350
Drug: Placebo — Oral 17 g dose of Placebo solution concentrate in a volume of approximately 30 mL, once a day, for 14 days.
  Arms: Placebo
Drug: Bisacodyl laxative tablets (rescue medication) — 5.0 mg tablets, 1 to 3 tablets in a single daily dose, to be provided for use as rescue medication if participant has not had bowel movement for 72 hours after start of treatment.

SUMMARY:
The purpose of this study is to compare the safety and tolerability of oral ingestion of PEG 3350 solution concentrate to oral ingestion of a placebo solution concentrate, in participants with constipation.

DETAILED DESCRIPTION:
This was a randomized, single-blind, placebo-controlled study to evaluate the proportion of participants with abnormalities of the oral mucosa detected by visual examination of the oral cavity in the polyethylene glycol (PEG) 3350 group compared with the placebo group. The study was also to evaluate the proportion of participants with abnormalities of the esophageal mucosa detected by endoscopic examination of the esophagus in the PEG 3350 group compared with the placebo group, and to compare the safety and tolerability by evaluation of the proportion of participants with the occurrence of adverse events (AEs) or adverse drug reactions.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory male or female with no history or current evidence of other conditions or abnormalities that would affect study results or interfere with participation for full duration of study
* meets diagnostic criteria for functional constipation. This includes loose stools that are rarely present without the use of laxatives and 2 or more of the following: straining during at least 25% of defecations; lumpy or hard stools in at least 25% of defecations; sensation of incomplete evacuation for at least 25% of defecations; sensation of anorectal obstruction/blockage for at least 25% of defecations; manual maneuvers to facilitate at least 25% of defecations [e.g., digital evacuation, support of the pelvic floor]; and fewer than 3 defecations per week. Criteria for functional constipation must be fulfilled for last 3 months, with symptom onset at least 6 months prior to diagnosis.
* continuous or recurrent symptoms for at least 3 months of: abdominal pain or discomfort, relieved with defecation, or associated with a change in frequency or consistency of stool, and an irregular pattern of defecation at least 25% of the time with 3 or more of the following: altered stool frequency, altered stool form (hard or loose/watery), altered stool passage (straining or urgency, feeling of incomplete evacuation), passage of mucus, and bloating or abdominal distension
* agrees to not use laxatives other than study medication for the duration of the study period
* agrees to not use disallowed concomitant medications for the duration of the study
* agrees to maintain a similar diet and level of activity from the period of the Screening Visit through End of Study
* individuals of reproductive potential must agree to remain abstinent or use (or have their partner use) 2 acceptable methods of birth control and until 2 weeks after the last dose of study drug in the last treatment period. Acceptable methods of birth control include: intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, condom, or vasectomy.

Exclusion Criteria:

* abnormal baseline endoscopy and/or an oral exam
* baseline oral exam showing evidence of oral lesions, such as herpes labialis or aphthous stomatitis, or known self-reported history or current periodontal gum disease
* history of impaired swallowing or difficulties swallowing foods and liquids
* known, history of, or suspected gastrointenstinal disease, including bowel perforation, obstruction, fecal impaction; irritable bowel syndrome (IBS), delayed gastric emptying, gastroparesis, gastroesophageal reflux disease (GERD), gastritis or peptic ulcer disease (PUD), dehydration, inflammatory bowel disease, bowel resection, anal fistulas/fissures, colostomy, etc.
* severe or unexplained abdominal pain
* history of or current alcohol or drug abuse
* history of malignancy ≤5 years prior to signing the informed consent, except for adequately treated basal cell and/or squamous cell skin cancer or in situ cervical cancer
* history of psychiatric illness requiring medications or hospitalization within the previous 12 months
* history of concurrent illness that required hospitalization within 4 weeks prior to Day -1 of the study
* allergies or allergic reactions or intolerance to any of the products used in study
* any degree of renal impairment
* major surgery or clinically significant illness within 4 weeks prior to Day -1 of Visit 1
* current or recent (within the past 30 days of signing informed consent) participation in a study with an investigational compound or device
* refusal to agree not to donate eggs or sperm upon the first study drug administration and thereafter through 90 days after the last study drug administration
* individual is an employee or family member of an employee of the sponsor or clinical unit where study will be conducted

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] McGraw T. Safety of polyethylene glycol 3350 solution in chronic constipation: randomized, placebo-controlled trial. Clin Exp Gastroenterol. 2016 Jul 15;9:173-80. doi: 10.2147/CEG.S111693. eCollection 2016. PMID 27486340

RESULTS

PARTICIPANT FLOW:
Groups:
- PEG 3350: Participants received a 17 g dose of PEG 3350 solution concentrate in a volume of approximately 30 mL, once a day, for 14 days. Bisacodyl laxative tablets, 5.0 mg, 1 to 3 tablets in a single daily dose, were provided for use as a rescue medication if a participant had not had a bowel movement for 72 hours after start of treatment.
- Placebo: Participants received a 17 g dose of Placebo solution concentrate solution in a volume of approximately 30 mL, once a day, for 14 days. Bisacodyl laxative tablets, 5.0 mg, 1 to 3 tablets in a single daily dose, were provided for use as a rescue medication if a participant had not had a bowel movement for 72 hours after start of treatment.
Period: Overall Study
Arm/Group | PEG 3350 | Placebo
Started | 31 | 34
Completed | 29 | 33
Not Completed | 2 | 1
Not completed — Withdrawal of Consent | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population, which consisted of all participants who received at least 1 dose of PEG 3350 or placebo and had at least 1 postdose safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | PEG 3350 | Placebo | Total
Number analyzed (Participants) | 31 | 34 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.5 (13.87) | 48.0 (15.17) | 46.4 (14.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 51
  Male | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Inflammation of the Oral Mucosa
Description: Participants underwent visual examination of the oral muscosa at Visit 2 and Visit 3. Measurements were based on 0-3 Likert Scale Scores: 0 = No inflammation (no erythema, no erosion/ulceration); 1 = Mild inflammation (erythema without erosion/ulceration); 2 = Moderate inflammation (erythema with erosion); 3 = Severe inflammation (erythema with ulceration).
Time Frame: Visit 2 (Day 1) and Visit 3 (Day 17 ± 2 days), up to 19 days after start of treatment
Population: as for baseline characteristics
Measure: Number; unit: Particpants
Arm/Group | PEG 3350 | Placebo
Number analyzed (Participants) | 31 | 34
Particpants
  Visit 2: 0=No inflammation | 31 | 34
  Visit 2: 1=Mild inflammation | 0 | 0
  Visit 2: 2=Moderate inflammation | 0 | 0
  Visit 2: 3=Severe inflammation | 0 | 0
  Visit 2: Not evaluated | 0 | 0
  Visit 3: 0=No inflammation | 29 | 33
  Visit 3: 1=Mild inflammation | 0 | 0
  Visit 3: 2=Moderate inflammation | 0 | 0
  Visit 3: 3=Severe inflammation | 0 | 0
  Visit 3: Not evaluated | 2 | 1

2. Primary Outcome: Number of Participants With Inflammation of the Esophageal Mucosa
Description: Participants underwent endoscopic examination of the esophageal mucosa at Visit 2 and Visit 3. Measurements were based on 0-3 Likert Scale Scores: 0 = No inflammation (no erythema, no erosion/ulceration); 1 = Mild inflammation (erythema without erosion/ulceration); 2 = Moderate inflammation (erythema with erosion); 3 = Severe inflammation (erythema with ulceration).
Time Frame: Visit 2 (Day 1) and Visit 3 (Day 17 ± 2 days), up to 19 days after start of treatment
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | PEG 3350 | Placebo
Number analyzed (Participants) | 31 | 34
Participants
  Visit 2: 0=No inflammation | 31 | 34
  Visit 2: 1=Mild inflammation | 0 | 0
  Visit 2: 2=Moderate inflammation | 0 | 0
  Visit 2: 3=Severe inflammation | 0 | 0
  Visit 2: Not evaluated | 0 | 0
  Visit 3: 0=No inflammation | 26 | 29
  Visit 3: 1=Mild inflammation | 2 | 1
  Visit 3: 2=Moderate inflammation | 1 | 3
  Visit 3: 3=Severe inflammation | 0 | 0
  Visit 3: Not evaluated | 2 | 1

ADVERSE EVENTS:
Time Frame: Up to 44 days after start of treatment
Arm/Group | PEG 3350 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/34
Other Adverse Events (participants affected / at risk) | 11/31 | 17/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG 3350 (N=31) | Placebo (N=34)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 6 (7)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 4 (4)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 2 (3)
Headache (Nervous system disorders) | 6 (8) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators have agreed to provide the Sponsor with the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication or presentation.